CLINICAL TRIAL: NCT07004764
Title: Enhancing Wound Perfusion in High-Risk Lower Extremity Orthopaedic Surgery: A Feasibility Study on Nitropaste Using Intraoperative SPY Imaging.
Brief Title: Enhancing Wound Perfusion in High-Risk Lower Extremity Orthopaedic Surgery: A Study on Nitropaste Using Intraoperative SPY Imaging.
Acronym: SPY NITROPASTE
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Orthopaedic Trauma Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00502503
Record Dates: First submitted 2025-05-27; First posted 2025-06-04 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Achilles Tendon Repairs/Reconstructions; Pilon Fracture of Tibia; Tibial Plateau Fracture; Ankle Fracture (Bimalleolar Equivalent, Bimalleolar, or Trimalleolar); Calcaneus Fractures; Talus Fracture; Wound Infection Deep; Wound Infection Post-Traumatic; Wound Dehiscence, Surgical
Keywords: Laser-assisted indocyanine green angiography; nitropaste; nitroglycerin; topical nitroglycerin; Achilles tendon repairs/reconstructions; Pilon Fracture of Tibia; Tibial Plateau Fracture; Ankle Fracture (bimalleolar equivalent, bimalleolar, or trimalleolar); Calcaneus Fractures; Talus fracture; Wound Dehiscence; Wound infection; tissue perfusion; Orthopaedic surgery
MeSH Terms: conditions — Tibial Plateau Fractures; Ankle Fractures; Surgical Wound Dehiscence; Wound Infection

STUDY DESIGN:
Intervention Model Description: This study is a single-arm open-label prospective clinical trial with no randomization or placebo. All patients will serve as own controls for LA-ICG fluorescence measurement. This study is considered a Phase I feasibility study, or a Stage 2a Development study under the IDEAL Framework
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nitropaste (Experimental): All patients enrolled in this study will receive a baseline perfusion measurement with the LA-ICG system. This will occur after wound closure. Subsequently, all patients will receive a single dose of nitropaste intraoperatively and a final LA-ICG tissue perfusion measurement.
  Interventions: Drug: Nitroglycerin Ointment 2%

INTERVENTIONS:
Drug: Nitroglycerin Ointment 2% — Patients will have pre- and post-nitropaste tissue perfusion measurement with the LA-ICG system.

SUMMARY:
Enhancing Wound Perfusion in High-Risk Lower Extremity Orthopaedic Surgery: A Feasibility Study on Nitropaste Using Intraoperative SPY Imaging.

DETAILED DESCRIPTION:
Tissue perfusion is a critical determinant of wound healing, particularly in lower extremity surgery where wound necrosis, dehiscence, and infection can result in limb loss. Despite current advances in wound therapy, rates of wound complications for certain lower extremity incisions remain high. Thus, there remains a critical need to identify agents that may potentially augment wound healing in orthopaedic surgery.

Nitropaste has been successfully used in plastic surgery to enhance perfusion and reduce flap necrosis, but its role in orthopaedic surgery is under-explored. In a meta-analysis of 6947 patients from 3 randomized controlled trials (RCTs) and 2 retrospective studies found that the use of nitropaste was associated with 0.23 odds [0.10-0.53, 95% confidence interval] of reduced mastectomy flap failure. Preliminary data from the investigator's institution involving 18 patients who received intraoperative nitropaste showed no adverse hypotensive effects, though wound complications occurred in three cases. Laser Assisted Indocyanine Green (LA-ICG) provides real-time, quantitative perfusion measurements, making it an ideal tool to evaluate the efficacy of nitropaste. Therefore, The purpose of this study is to evaluate the effects of nitropaste on immediate tissue perfusion and wound complications in high-risk lower extremity orthopaedic incisions using LA-ICG. Additionally, the investigators will assess the safety of single-dose nitropaste in these patients. The investigators hypothesize that intraoperative nitropaste application will significantly improve tissue perfusion, which in turn would be associated with reduced wound complications, with minimal adverse effects.

Aim 1: To evaluate the effect of nitropaste on immediate tissue perfusion in lower extremity orthopaedic incisions using LA-ICG.

1. Primary outcomes: Relative fluorescence unit (RFU), absolute fluorescence units (AFU), mean incision perfusion (MIP), and mean perfusion impairment (MPI)
2. Null hypothesis: The investigators hypothesize that nitropaste would not be associated with a significant increase in perfusion, as measured by RFU, AFU, MIP and MPI.

Aim 2: To assess trial feasibility and ability to identify wound complications for a future large-scale trial.

1. Primary outcomes: Recruitment rate, retention rate, and wound complications, which include wound dehiscence, wound necrosis, superficial infection, and deep infection.
2. Recruitment goal: 50% recruitment at 8 months
3. Retention rate goal: 80% of patients with minimum of 3 months follow-up at trial conclusion
4. No a priori hypotheses.

Aim 3: To assess the safety of nitropaste in lower extremity orthopaedic surgeries.

1. Secondary outcomes: Hypotension, headache, dizziness, allergic reactions, and other adverse events.
2. No a priori hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Undergoing surgery for one of the following procedures:

  * Current Procedural Terminology (CPT) 28415 - Open reduction calcaneal fracture ± internal/external fixation
  * CPT-27814 - Open reduction of bimalleolar fracture ± internal/external fixation
  * CPT-27822 - Open reduction trimalleolar ankle fracture, medial and lateral malleoli only, ± internal/external fix
  * CPT-27823 - Open reduction trimalleolar ankle fracture, including posterior malleolus, ± internal/external fix
  * CPT-27826 - Open reduction pilon fracture, internal/external fixation of fibula ONLY
  * CPT-27827 - Open reduction pilon fracture, internal/external fixation of tibia ONLY
  * CPT-27828 - Open reduction pilon fracture, internal/external fixation of tibia AND fibula
  * CPT-27535 - Open reduction unicondylar tibial plateau fracture, ± internal/external fixation
  * CPT-27536 - Open reduction bicondylar tibial plateau fracture, ± internal/external fixation
  * CPT-28445 - Open reduction of talus fracture, ± internal/external fixation
  * CPT-27650 - Primary Achilles tendon repair
* English-speaking
* Able to provide informed consent during preoperative clinic visit, in the preoperative nursing area, or on inpatient units.

Exclusion Criteria:

* Contraindications to nitroglycerin, including known allergy.
* Allergy to indocyanine green or components of ICG dye, including allergies to iodine or shell-fish.
* Severe kidney injury, as determined by attending surgeon and/or anesthesiologist, that would impair clearance of ICG dye.
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Absolute fluorescence unit (AFU) | Intraoperative measurement
  raw fluorescence measurement
Relative fluorescence unit (RFU) | Intraoperative measurement
  Will be calculated as a ratio of the mean fluorescence measure to the mean "normal" measurement. The mean "normal" measurement will be defined as the maximal signal intensity in a region outside of the wound area.
mean incision perfusion (MIP) | Intraoperative measurement
  the mean fluorescence of 10 points adjacent to the incision.
mean perfusion impairment (MPI) | Intraoperative measurement
  the difference between mean of each pair of points on each side of the incision.

SECONDARY OUTCOMES:
Number of Participants with Wound dehiscence | From surgery to 3 months post-operation
  participants with wound dehiscence (when two edges of a wound separate)
Number of participants with Wound necrosis | From surgery to 3 months post-operation
  participants with any death of peri-incisional skin
Number of participants with Superficial infection | From surgery to 3 months post-operation
  participants with any wound infection that is treated only with oral antibiotics
Number of participants with Deep infection | From surgery to 3 months post-operation
  Any wound infection that requires surgical management

OTHER OUTCOMES:
recruitment rate | From study start to final recruitment approximately 8 months
  Patients recruited into the study per time and per patients approached
retention rate | From study start to 3 months after final patient is recruited
  Percent patient follow-up at 3 months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Henry T Shu, MD, Study Director — Johns Hopkins University; Babar Shafi, MD, MSPT, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No
No sharing will occur to protect patient Protected Health Information (PHI)

REFERENCES:
- [Background] Sanniec K, Teotia S, Amirlak B. Management of Tissue Ischemia in Mastectomy Skin Flaps: Algorithm Integrating SPY Angiography and Topical Nitroglycerin. Plast Reconstr Surg Glob Open. 2016 Oct 6;4(10):e1075. doi: 10.1097/GOX.0000000000001075. eCollection 2016 Oct. PMID 27826472